CLINICAL TRIAL: NCT04736134
Title: A Double-blind, Placebo-controlled, Randomized, Single and Multiple Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous and Subcutaneous Administration of BMS-986326 in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, Drug Levels, and Drug Effects of BMS-986326 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM034-001; 2020-002763-64 (EudraCT Number); U1111-1252-7566 (Registry Identifier: WHO)
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Healthy Participants
Keywords: BMS-986326; Healthy participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Active Treatment (BMS 986326) IV (Experimental): Intravenous (IV)
  Interventions: Biological: BMS-986326
- Active Treatment (BMS 986326) SC (Experimental): Subcutaneous (SC)
  Interventions: Biological: BMS-986326
- Placebo IV (Placebo Comparator)
  Interventions: Other: Placebo matching BMS-986326
- Placebo SC (Placebo Comparator)
  Interventions: Other: Placebo matching BMS-986326
- Multiple Ascending Dose Placebo SC (Placebo Comparator): Placebo
  Interventions: Other: Multiple Ascending Dose Placebo
- Multiple Ascending Dose SC (Experimental): BMS 986326 SC
  Interventions: Biological: Multiple Ascending Dose SC

INTERVENTIONS:
Biological: BMS-986326 — Specified dose on specified days
  Arms: Active Treatment (BMS 986326) IV; Active Treatment (BMS 986326) SC
Other: Placebo matching BMS-986326 — Specified dose on specified days
  Arms: Placebo IV; Placebo SC
Biological: Multiple Ascending Dose SC — Specified dose on specified days
  Arms: Multiple Ascending Dose SC
Other: Multiple Ascending Dose Placebo — Specified dose on specified days
  Arms: Multiple Ascending Dose Placebo SC

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, drug levels, drug effects, and immunogenicity of BMS-986326 after infusion or injection in healthy participants. The results of this study will guide the selection of the dose range, dosing frequency, and the route of administration for future studies of BMS-986326 in participants with immune-mediated diseases.

ELIGIBILITY:
Inclusion Criteria:

* In good health, as determined by the investigator based on a physical examination at screening
* Body mass index (BMI) ≥ 18 and ≤ 30 kg/m^2 at screening
* Afebrile, with supine systolic blood pressure (BP) ≥ 90 and ≤ 140 mmHg and supine diastolic BP ≥ 50 and ≤ 90 mmHg and heart rate ≥ 50 and ≤ 90 bpm at screening
* Male participants are eligible to participate in cohorts (A1-B3).Women not of child bearing potential (WNOCBP) are eligible to participate in all cohorts (A1-B3 and C1-C2) Women of child-bearing potential (WOCBP) are only eligible for the subcutaneous (SC) cohorts (B1-B3 and C1-C2)
* Must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Women who are pregnant or lactating
* History of, or active, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, echocardiogram (ECG), or clinical laboratory determinations beyond what is consistent with healthy participants
* History of serious adverse reaction or hypersensitivity to any (subcutaneous) SC- or (intravenous) IV-administered biological therapeutic, including IV immunoglobulins and human blood products

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 175 days
Number of participants with clinical laboratory abnormalities | Up to 175 days
Number of participants with vital sign abnormalities | Up to 175 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 175 days
Number of participants with physical examinations abnormalities | Up to 175 days

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Up to 175 days
Time of maximum observed serum concentration (Tmax) | Up to 175 days
Area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] | Up to 175 days
Geometric mean ratios of test (SC) vs reference (IV): Area under the serum concentration-time curve extrapolated to infinite time [AUC(INF)] | Up to 175 days
Change in regulatory T cells (Treg) count | Up to 175 days
Change in Treg-to-conventional CD4 cells [Treg-to-Tconv] ratio | Up to 175 days
Number of participants with anti-drug antibodies | Up to 175 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Berlin, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome